CLINICAL TRIAL: NCT03273257
Title: A Phase 2, Randomised, Double-Blind, Placebo-Controlled, Multicentre, Prospective Study to Assess Efficacy of Riociguat in Patients With Operable CTEPH Prior to Pulmonary Endarterectomy With High Preoperative Pulmonary Vascular Resistance
Brief Title: Riociguat in Patients With Operable CTEPH Prior to Pulmonary Endarterectomy (PEA Bridging Study)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to slower than expected recruitment and the additional limitations on clinical research imposed by the COVID-19 pandemic, both of which made study completion within a reasonable timeframe appear unlikely.
Sponsor: International CTEPH Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEA Bridging Study
Record Dates: First submitted 2017-08-25; First posted 2017-09-06 (Actual); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; CTEPH
Keywords: Pulmonary endarterectomy; PEA; Medical therapy
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riociguat (Active Comparator): Patients will receive riociguat for 3 months followed by pulmonary endarterectomy.
  Interventions: Drug: Riociguat; Procedure: Pulmonary endarterectomy
- Placebo (Placebo Comparator): Patients will receive placebo for 3 months followed by pulmonary endarterectomy.
  Interventions: Drug: Placebo; Procedure: Pulmonary endarterectomy

INTERVENTIONS:
Drug: Riociguat — Riociguat will be initiated at 1 mg tid. The dosage will be increased by 0.5 mg at 2 week intervals based on tolerability as assessed by systolic blood pressure up to a maximum dose of 2.5 mg tid.
  Downtitration to 0.5 mg tid is foreseen for patients with low optimal tolerability.
  Other Names: Adempas; BAY 63-2521
  Arms: Riociguat
Drug: Placebo — Placebo will be given analogue to riociguat with matching tablets.
  Arms: Placebo
Procedure: Pulmonary endarterectomy — PEA will be performed at the end of medical treatment (Day 90)
  Other Names: PEA

SUMMARY:
This is a randomised, double-blind, placebo-controlled, multicentre, multinational, prospective study in patients with operable chronic thromboembolic pulmonary hypertension (CTEPH) prior to pulmonary endarterectomy (PEA) with high preoperative pulmonary vascular resistance (PVR). Patients will be randomised in a 1:1 ratio to receive riociguat or matching placebo for 3 months before undergoing PEA. The primary objective of this study is to assess the efficacy of riociguat on preoperative PVR compared to placebo in patients with operable CTEPH.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or nonpregnant and nonlactating female patient aged from 18 to 80 years, both inclusive
* Is diagnosed with operable CTEPH and anticipating symptomatic and/or prognostic benefit from PEA
* Has pulmonary vascular resistance (PVR) >800 dyn·s·cm-5
* Has undergone right heart catheterisation not more than 180 days before randomisation visit
* Has been treated with anticoagulants for at least 90 days before randomisation visit
* Has ability to swallow oral medication
* Has ability and willingness to participate and access the health facility
* Is capable of understanding the written informed consent and provides signed and witnessed written informed consent
* Female patient must be either surgically sterile, postmenopausal (no menses for the previous 12 months), or must be practicing an effective method of birth control as determined by the investigator (eg, oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or male partner with vasectomy or complete abstinence)

Exclusion Criteria:

* Has unstable disease in need of urgent PEA surgery as determined by the treating physician
* Has known hypersensitivity, allergic, or adverse reactions to riociguat or any of the excipients comprising riociguat tablets.
* Has known active hepatitis A IgM (HAV-IgM), hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV Ab)
* Is human immunodeficiency virus positive
* Has pulmonary veno-occlusive disease
* Has symptomatic hypotension
* Has symptomatic carotid disease
* Has significant coronary atherosclerotic disease in need of intervention
* Has severe left heart disease in need of intervention
* Has redo sternotomy
* Has received any background therapy for pulmonary arterial hypertension (PAH) in the preceding 30 days before randomisation visit including endothelin receptor antagonists (ERAs), phosphodiesterase 5 (PDE5) inhibitors, or prostanoids
* Is receiving nitrates, nitric oxide donors (e.g. amyl nitrite), ERAs, prostanoids, specific PDE5 inhibitors, nonspecific phosphodiesterase inhibitors (e.g. dipyridamole, theophylline)
* Is receiving strong cytochrome P450 (CYP) and P-glycoprotein/breast cancer resistance protein inhibitors
* Is receiving strong CYP3A inducers
* Has creatinine clearance <15 mL/min or on any form of dialysis
* Has severe hepatic impairment classified as Child-Pugh C
* Has received an investigational drug within the past 4 weeks before randomisation visit
* Is a lactating or pregnant (as demonstrated by a serum pregnancy test) woman, and not willing to take measures for not to become pregnant during the 3 months treatment study period and one month after the last dose of study drug administered
* Has smoked or used tobacco in any form, including snuff or chewing within 3 months prior to randomisation visit
* Has idiopathic interstitial pneumonitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jenkins, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust, Cambridge, UK
Locations (4):
- UC San Diego, La Jolla, California, United States
- Hopital de Bicêtre, Paris, France
- Kerckhoff-Klinik GmbH, Bad Nauheim, Germany
- Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not foreseen

REFERENCES:
- See also: Website of the International CTEPH Association — https://www.cteph-association.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were recruited at 3 expert centers for CTEPH in France, Germany and the UK between August 2018 and May 2020.
Groups:
- Riociguat: Patients will receive riociguat for 3 months followed by pulmonary endarterectomy.
  Riociguat will be initiated at 1 mg tid. The dosage will be increased by 0.5 mg at 2 week intervals based on tolerability as assessed by systolic blood pressure up to a maximum dose of 2.5 mg tid.
  Downtitration to 0.5 mg tid is foreseen for patients with low optimal tolerability.
  PEA will be performed at the end of medical treatment (Day 90)
- Placebo: Patients will receive placebo for 3 months followed by pulmonary endarterectomy.
  Placebo will be given analogue to riociguat with matching tablets.
  PEA will be performed at the end of medical treatment (Day 90)
Period: Overall Study
Arm/Group | Riociguat | Placebo
Started | 7 | 7
Started Treatment | 7 | 6 (Only 6 patients from the placebo group started treatment because 1 patient died after randomization (= study start), but before initiating treatment)
Underwent PEA | 6 | 5
Completed | 3 | 3
Not Completed | 4 | 4
Not completed — Death | 0 | 1
Not completed — Inability to schedule PEA according to the protocol due to the COVID pandemic | 1 | 1
Not completed — Study terminated | 3 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of randomized study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Median (Full Range); unit: years] | 66 [48 to 75] | 67 [52 to 74] | 66 [48 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 31.2 (3.9) | 25.4 (1.7) | 28.8 (4.3)
PVR at diagnosis [Mean (Standard Deviation); unit: dyn*sec/cm^5] | 944.0 (92.7) | 1007.5 (368.2) | 973.3 (248.8)
Mean pulmonary arterial pressure (mPAP) at diagnosis [Mean (Standard Deviation); unit: mmHg] | 50.3 (8.4) | 53.2 (4.8) | 51.5 (7.0)
Received beta blockers between enrollment and PEA [Count of Participants; unit: Participants] | 3 | 0 | 3
Received vitamin K antagonists between enrollment and PEA [Count of Participants; unit: Participants] | 1 | 2 | 3
Received new/direct oral anticoagulants between enrollment and PEA [Count of Participants; unit: Participants] | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) to Immediately Before Pulmonary Endarterectomy (Pre-PEA)
Description: Pulmonary vascular resistance (PVR) will be assessed at baseline and immediately before pulmonary endarterectomy. The change in PVR will be assessed as percentage.
Time Frame: 90 days
Population: All participants who received at least one dose of randomized study drug and underwent PEA before study termination
Measure: Mean (Standard Deviation); unit: percentage of baseline PVR
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 6 | 5
percentage of baseline PVR | -28.4 (16.2) | -6.9 (27.9)
Statistical Analysis 1: Comparison: Riociguat vs Placebo; The null hypothesis is that there is no difference between the treatment groups in percent change from baseline in PVR immediately before PEA; Test type: Superiority; p = 0.139, 2-sample Wilcoxon rank sum test

2. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) to 6 Months Post Pulmonary Endarterectomy (PEA)
Description: Pulmonary vascular resistance (PVR) will be assessed at baseline and 6 months post pulmonary endarterectomy (PEA). The change in PVR will be assessed as percentage.
Time Frame: 270 days
Population: All participants who received at least one dose of randomized study drug and completed the study prior to study termination
Measure: Mean (Standard Deviation); unit: percentage of baseline PVR
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 3 | 3
percentage of baseline PVR | -68.1 (9.8) | -83.0 (2.2)

3. Secondary Outcome: Number of Patients With Either All-cause Death, PH-related Hospitalization, Need for PAH-targeted Therapy or WHO Functional Class Unchanged or Worse Between Randomization and 6 Months Post Pulmonary Endarterectomy (Composite Endpoint)
Description: All deaths occurring post-randomization until the last visit will be included. All PH-related hospitalizations except the in-hospital care during and after pulmonary endarterectomy (PEA) from randomization until 6 months after PEA will be included.
  The worst value for World Health Organization (WHO) functional class after treatment will be used.
Time Frame: 270 days
Population: All participants who underwent PEA before study termination
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 6 | 5

4. Secondary Outcome: Intraoperative Circulatory Arrest Time
Description: Circulatory arrest time will be measured in minutes
Time Frame: intraoperative
Population: All participants who underwent PEA before study termination
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 6 | 5
minutes | 32 (9) | 40 (12)

5. Secondary Outcome: Number of Patients With Intraoperative Surgery-related Complications (Composite Endpoint)
Description: The occurrence of any of the following complications will be assessed:
  * Bleeding and/or blood loss >1 L in 12 hours
  * Airway bleed with need for extracorporeal membrane oxygenation
  * Any use of extracorporeal membrane oxygenation for respiratory or hemodynamic support, specified as veno-venous or veno-arterial
  * Prolonged ventilation >96 hours
  * Need for tracheostomy
  * Need for drainage of pericardial effusion
  * Neurological complications, ie, stroke, cerebral, subdural bleeding
  * Reintubation or noninvasive ventilation for reperfusion response
  * Hemoptysis requiring any intervention
  * Renal failure requiring dialysis
  * Wound infections
  * Pneumonia
  * Prolonged need for inotropic support (≥ 5 days)
Time Frame: intraoperative
Population: All participants who underwent PEA before study termination
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

6. Secondary Outcome: Surgical Evaluation of Specimen: Stratification of Patients According to Ease of Dissection Plane
Description: Classed as easier than normal (1); normal (2); more difficult than normal (3)
Time Frame: intraoperative
Population: All participants who underwent PEA
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Easier than normal | 1 | 1
  Normal | 3 | 4
  More difficult than normal | 2 | 0

7. Secondary Outcome: Surgical Evaluation of Specimen: Stratification of Patients According to Completeness of Disease Clearance
Description: Classed as better than expected (1); as expected (2); worse than expected (3)
Time Frame: intraoperative
Population: All participants who underwent PEA before study termination
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Better than expected | 0 | 0
  As expected | 6 | 5
  Worse than expected | 0 | 0

8. Secondary Outcome: Surgical Evaluation of Specimen: Stratification of Patients According to Appearance of Clot and Vessel Wall
Description: Classed as more solid than usual (1); normal (2); more friable than usual (3)
Time Frame: intraoperative
Population: All participants who underwent PEA before study termination
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  More solid than usual | 0 | 0
  Normal | 4 | 5
  More friable than usual | 2 | 0

9. Secondary Outcome: Number of Patients Who Died During the Course of the Study
Description: All deaths occurring during the whole course of the study
Time Frame: 270 days
Population: All participants who underwent PEA before study termination
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

10. Secondary Outcome: Patients Who Withdraw During the Randomized Treatment Phase
Description: Only withdrawals after randomization but before PEA will be included
Time Frame: 90 days
Population: All participants who received at least one dose of randomized study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 7 | 6
Participants | 1 | 1

11. Other Pre Specified Outcome: Change in NT-proBNP From Baseline Until the End of Medical Treatment
Description: Data are not reported for this exploratory endpoint because of limited sample size due to early termination of the study
Time Frame: 90 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in NT-proBNP From Baseline Until 6 Months Post-surgery
Description: as for outcome 11
Time Frame: 270 days
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Cardiac Index From Baseline Until the End of Medical Treatment
Description: as for outcome 11
Time Frame: 90 days
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Cardiac Index From Baseline Until 6 Months Post-surgery
Description: as for outcome 11
Time Frame: 270 days
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Mean Right Atrial Pressure From Baseline Until the End of Medical Treatment
Description: as for outcome 11
Time Frame: 90 days
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Mean Right Atrial Pressure From Baseline Until 6 Months Post-surgery
Description: as for outcome 11
Time Frame: 270 days
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Mean Pulmonary Atrial Pressure From Baseline Until the End of Medical Treatment
Description: as for outcome 11
Time Frame: 90 days
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Mean Pulmonary Atrial Pressure From Baseline Until 6 Months Post-surgery
Description: as for outcome 11
Time Frame: 270 days
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Pulmonary Artery Wedge Pressure From Baseline Until the End of Medical Treatment
Description: as for outcome 11
Time Frame: 90 days
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Pulmonary Artery Wedge Pressure From Baseline Until 6 Months Post-surgery
Description: as for outcome 11
Time Frame: 270 days
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Length of Hospital Stay for Pulmonary Endarterectomy
Description: as for outcome 11
Time Frame: intraoperative
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Length of Intensive Care Unit Stay for Pulmonary Endarterectomy
Description: as for outcome 11
Time Frame: intraoperative
Reporting Status: Not Posted

23. Other Pre Specified Outcome: WHO Functional Class at the End of Medical Treatment
Description: as for outcome 11
Time Frame: 90 days
Reporting Status: Not Posted

24. Other Pre Specified Outcome: WHO Functional Class 6 Months Post Pulmonary Endarterectomy
Description: as for outcome 11
Time Frame: 270 days
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Need for PAH-targeted Therapy 6 Months Post-surgery
Description: as for outcome 11
Time Frame: 270 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From informed consent until study completion (typically 9-12 months) or early termination
Description: Events reported are treatment-emergent adverse events, i.e. any event not present before exposure to study drug or any event already present that worsened in either intensity or frequency after exposure to study drug, in patients who actually received any study drug. Events were identified by investigator assessment at each visit, and from study data. All-cause mortality is reported based on all patients enrolled, including one patient who died prior to initiating treatment.
Groups:
- Riociguat: Patients will receive riociguat for 3 months followed by pulmonary endarterectomy.
  Riociguat will be initiated at 1 mg. The dosage will be increased by 0.5 mg at 2 week intervals based on tolerability as assessed by systolic blood pressure up to a maximum dose of 2.5 mg tid.
  Downtitration to 0.5 mg tid is foreseen for patients with low optimal tolerability.
  PEA will be performed at the end of medical treatment (Day 90)
Arm/Group | Riociguat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/7
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/6
Other Adverse Events (participants affected / at risk) | 7/7 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (N=7) | Placebo (N=6)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Worsening symptoms of CTEPH, including increased NT-proBNP, peripheral oedema and breathlessness
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (N=7) | Placebo (N=6)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (4)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug therapy (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated after enrolling only 14 out of 88 planned patients, due to slower than expected recruitment and the additional limitations on clinical research imposed by the COVID-19 pandemic. No firm conclusions can be drawn based on the study data due to the limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Both the International CTEPH Association and the financial sponsor can review results communications prior to public release and can embargo communications regarding trial results for up to 180 days from submission for review

DOCUMENTS (2):
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT03273257/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT03273257/SAP_001.pdf